CLINICAL TRIAL: NCT03427502
Title: Anterior Ethmoidal Nerve Block in Prevention of Postoperative Agitation Following Nasal Surgeries With Nasal Packs Under General Anesthesia: A Double Blind Randomized Control Trial
Brief Title: Anterior Ethmoidal Nerve Block in Prevention of Postoperative Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumbini Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 139
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Agitation: Impaired Awareness, Abnormal Cognitive Function, Confusion, and Verbal and Physical Agitation During Recovery From General Anesthesia; Deviated Nasal Septum; Chronic Rhinosinusitis (Diagnosis); Nasal Polyps
Keywords: general anesthesia; nasal surgery; anterior ehtmoidal nerve block; bupivacaine; postoperative confusion
MeSH Terms: conditions — Confusion; Disease; Nasal Polyps | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Experimental: Study Group At the end of surgery before nasal packing, scrub nurse will prepare 10 ml solution 0.5% bupivacaine with 1:2,00,000 adrenaline in a syringe and pass it over to the operating surgeon. The surgeon will block anterior ethmoidal nerve.
  Injection technique: External nasal nerve will be blocked through an inter-cartilaginous injection into the dorsum of the nose.
  Internal nasal nerve will be blocked in septum and lateral wall of nose. Septal block is done in upper anterior part of nasal septum. Three injections will be given on lateral nasal wall. First injection will be given just antero-superior to the attachment of middle turbinate (axilla). Second injection will be given at the anterior end of middle turbinate and third injection at the medial surface of middle turbinate. Withdrawal of injection will be done prior to deposition of solution every time to ensure that the solution is not deposited directly into a blood vessel.
  Interventions: Drug: Bupivacaine-epinephrine
- Control Group (Placebo Comparator): At the end of surgery before nasal packing, scrub nurse will pass 10 ml of normal saline in a syringe to the surgeron.
  Injection technique remains the same as in Study group.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — 10 ml of 0.5% bupivacaine with 1:2,00,000 adrenaline. For children less than 12 years of age, 0.25% bupivacaine with 1:2,00,000 adrenaline
  Arms: Study Group
Drug: normal saline — normal saline
  Arms: Control Group

SUMMARY:
Postoperative agitation is an important complication of general anesthesia, moreover, it has been found with high incidence in ear, nose, throat (ENT) surgeries. We aim to study whether anterior ethmoidal nerve block will be successful in reducing postoperative agitation in those patients. Study population will be randomized into two groups, treatment and control group. Anterior ethmoidal nerve block will be done in treatment group and postoperative agitation compared between these two groups. Agitation score will be scored with Riker Sedation-Agitation Scale (SAS).

Ho: Occurrence of post-operative agitation in patients undergoing nasal surgery with nasal pack under general anesthesia is equal in those with ethmoidal nerve block as compared to those without the block.

Ha: Occurrence of post-operative agitation in patients undergoing nasal surgery with nasal pack under general anesthesia is not equal in those with ethmoidal nerve block as compared to those without the block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing nasal surgery
* Under General Anesthesia
* With nasal packs

Exclusion Criteria:

* Do not consent to the study.
* History of allergy to lignocaine or bupivacaine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative agitation | After extubation before leaving operation table, an average of 10 minutes
  It will be assessed with Riker Sedation-Agitation Scale (SAS). It is a Likert scale with scores from 1 to 7 where 1 indicates unarousable (Minimal or no response to noxious stimuli, does not communicate or follow commands) and 7 indicates Dangerous agitation (Pulling at ET tube, trying to remove catheters, climbing over bedrail, striking at staff, thrashing side-to-side). A higher value indicates worse outcome.
Postoperative agitation | 30 minutes after first score.
  It will be assessed with Riker Sedation-Agitation Scale (SAS). It is a Likert scale with scores from 1 to 7 where 1 indicates unarousable (Minimal or no response to noxious stimuli, does not communicate or follow commands) and 7 indicates Dangerous agitation (Pulling at ET tube, trying to remove catheters, climbing over bedrail, striking at staff, thrashing side-to-side). A higher value indicates worse outcome.
Postoperative agitation | 9:00 AM next morning
  It will be assessed with Riker Sedation-Agitation Scale (SAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Lumbini Medical College, Tānsen, Palpa, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
All data except patients name and address may be shared.